CLINICAL TRIAL: NCT02491151
Title: Fluconazole Exposure in Critically Ill Patients and the Value of Therapeutic Drug Monitoring
Brief Title: Variability of Fluconazole Concentration in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, Associate Professor of Medicine, University Medical Center Groningen
Other Study IDs: FLU-14O28
Record Dates: First submitted 2015-06-17; First posted 2015-07-07 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Invasive Candidiasis
MeSH Terms: conditions — Candidiasis, Invasive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Fluconazole is the first-line agent in the treatment of invasive candidiasis. Studies showed inappropriate drug exposure causes high mortality in critically ill patients. Under-dosing and ineffective fluconazole trough serum concentrations were found in a recent retrospective study. Variability in fluconazole exposure can be easily measured with therapeutic drug monitoring. For patient groups who are at risk for drug underexposure, therapeutic drug monitoring can be valuable regards decreasing mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older.
* Treatment with fluconazole.
* Written informed consent obtained from patient.
* Written informed consent obtained from representative of patient.

Exclusion Criteria:

* Blood sampling not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the University Medical Center Groningen who receive fluconazole
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of fluconazole in critically ill patients | Up to one month
  Plasma concentrations of fluconazole will be determined using a validated method involving LC-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Jan-WIllem Alffenaar, PharmD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Boonstra JM, Martson AG, Sandaradura I, Kosterink JGW, van der Werf TS, Marriott DJE, Zijlstra JG, Touw DJ, Alffenaar JWC. Optimization of Fluconazole Dosing for the Prevention and Treatment of Invasive Candidiasis Based on the Pharmacokinetics of Fluconazole in Critically Ill Patients. Antimicrob Agents Chemother. 2021 Feb 17;65(3):e01554-20. doi: 10.1128/AAC.01554-20. Print 2021 Feb 17. PMID 33361296